CLINICAL TRIAL: NCT06680557
Title: Effects of Different Types of Exercises on Postprandial Blood Glucose Levels in Children and Adolescents With Type 1 Diabetes Mellitus
Brief Title: Exercises on Children and Adolescents With Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marina Safwat Ibrahim, Pediatric resident at Sohag University Hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-15-10__2MS
Record Dates: First submitted 2024-11-02; First posted 2024-11-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Each participant will be assigned to perform either the aerobic or the resistance exercise sessions following the lunch meal in a random sequence by the withdrawal of a sealed envelope containing a paper with a written random sequence of the two exercise sessions.
  The envelope will be withdrawn randomly and opened immediately before the first exercise session.
  The other type of exercise session will be performed after 48 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children and adolescents aged 10-18 years, diagnosed with T1DM for at least 1 year (Experimental): Each participant will be assigned to perform either the aerobic or the resistance exercise sessions following the lunch meal in a random sequence by the withdrawal of a sealed envelope containing a paper with a written random sequence of the two exercise sessions. The envelope will be withdrawn randomly and opened immediately before the first exercise session. The other type of exercise session will be performed after 48 hours.
  Interventions: Behavioral: Aerobic and resistance exercises

INTERVENTIONS:
Behavioral: Aerobic and resistance exercises — * Aerobic exercise session: A 30-minutes of brisk walking exercise on an indoor track without speed walking or running .
  * Resistant exercise session: A 30-minutes of resistance exercise using rubber bands including warm-up and cool-down periods. Rubber band exercises are composed of seven exercises: squat, leg extension, pull apart, seated row, standing biceps curl, overhead press and lateral raise. Each exercise consists of three sets of 10 repetitions with 1 minute rest between each exercise set.

SUMMARY:
This study aimed to assess the effect of aerobic and resistance exercise on postprandial blood glucose levels in children and adolescents aged 10 - 18 years, diagnosed with type 1 diabetes mellitus (T1DM) for at least 1 year, attending the Pediatric diabetes clinic at Sohag University Hospital and using multiple daily insulin (MDI) regimen.

DETAILED DESCRIPTION:
The participants will be admitted at the pediatric department, Sohag University Hospital for 1 week. Full history taking, thorough clinical examination, review of participants' medical files and assessment of their basal insulin doses ,Insulin to carbohydrate ratio(ICR) and Insulin sensitivity factor (ISF) will be done if required. During hospitalization, the study participants will be familiarized with the types of the exercises used and how to perform each exercise carefully with the help of an exercise specialist before the experimental sessions. The pre-exercise lunch meal will be standardized to provide 30% of the total daily caloric requirement for the study participant (50% carbohydrate, 30% fat and 20% protein). The meal will consist of rice, chicken breast, vegetables and fruits. The Lunch meals will be consumed at the pediatric department, Sohag university hospital at 2 PM. The meal will be consumed within 20 minutes. Each participant will be assigned to perform either the aerobic or the resistance exercise sessions following the lunch meal in a random sequence by the withdrawal of a sealed envelope containing a paper with a written random sequence of the two exercise sessions. The envelope will be withdrawn randomly and opened immediately before the first exercise session. The other type of exercise session will be performed after 48 hours.

Participants will wear a bracelet heart rate monitor during the exercise sessions. Each participant will perform each of the following 2 exercise sessions 30 minutes after the lunch meal in a random sequence with 48-hour period between the 2 exercise sessions

* Aerobic exercise session: A 30-minutes of brisk walking exercise on an indoor track without speed walking or running .
* Resistant exercise session: A 30-minutes of resistance exercise using rubber bands including warm-up and cool-down periods. Rubber band exercises are composed of seven exercises: squat, leg extension, pull apart, seated row, standing biceps curl, overhead press and lateral raise. Each exercise consists of three sets of 10 repetitions with 1 minute rest between each exercise set.

Following the exercise session, participants will be allowed to perform only sedentary activities. No food or drink - except water - will be allowed for the following 5 hours unless needed to correct hypoglycemia.

The participants will be instructed to avoid exercise the day before and on the same day of the experimental session. Capillary blood glucose level measured by a calibrated finger-prick blood glucose meter before the meal , immediately prior to exercise (30 minutes before the start of the meal), after the exercise (60 minutes after the start of the meal) and then every hour throughout the 6-hour postprandial period.

The blood glucose excursion throughout the 6-hour postprandial period is the primary outcome measure of the study. Secondary outcome measures included the time to peak and time to lowest blood glucose levels, blood glucose area under the curve (AUC) and the frequency of postprandial hypoglycemia among the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 10 - 18 years, diagnosed with T1DM for at least 1 year

Exclusion Criteria:

* Children and adolescents with associated diseases such as autoimmune hypothyroidism or celiac disease and those with diabetes-related complications such as diabetic neuropathy, retinopathy or nephropathy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
The blood glucose excursion throughout the 6-hour postprandial period. | Before the meal, immediately prior to exercise (30 minutes after the start of the meal), after the exercise (60 minutes after the start of the meal) and then every hour throughout the 6-hour postprandial period.
  Capillary blood glucose level measured by a calibrated finger-prick blood glucose meter.

SECONDARY OUTCOMES:
Blood glucose area under the curve (AUC) | 6 hours after the meal.
  Capillary blood glucose level measured by a calibrated finger-prick blood glucose meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided